CLINICAL TRIAL: NCT04277260
Title: Study on the Molecular Structure and Content of Human Milk Oligosaccharides (HMOs) in Breast Milk and Its Effect on Infant Health in China
Brief Title: Molecular Structure and Content of Human Milk Oligosaccharides (HMOs) and Its Effect on Infant Health in China
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Heilongjiang Feihe Dairy Co. Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: SCMCIRB-K2019023-2
Record Dates: First submitted 2020-02-13; First posted 2020-02-20 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Child Development

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Fecal specimen of infants
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Full term delivery: In the cooperative obstetric hospital, 30 cases of full-term delivery healthy mothers and their infants are selected. Each pair of nursing mothers and infants will complete the observation for 6 months. The samples of human milk and newborn feces are the experimental objects.
- Preterm delivery(35-37 weeks): In the cooperative obstetric hospital, 30 cases of preterm delivery(35-37 weeks) mothers and their infants are selected. Each pair of nursing mothers and infants will complete the observation for 6 months. The samples of human milk and newborn feces are the experimental objects.
- Preterm delivery(32-35 weeks): In the cooperative obstetric hospital, 30 cases of preterm delivery(32-35 weeks) mothers and their infants are selected. Each pair of nursing mothers and infants will complete the observation for 6 months. The samples of human milk and newborn feces are the experimental objects.
- Preterm delivery(28-32 weeks): In the cooperative obstetric hospital, 30 cases of preterm delivery(28-32 weeks) mothers and their infants are selected. Each pair of nursing mothers and infants will complete the observation for 6 months. The samples of human milk and newborn feces are the experimental objects.

SUMMARY:
In the study, the composition and content of human milk oligosaccharides in premature delivery mothers in China will be examined to investigate the differences in oligosaccharide concentrations in preterm breast milk from different gestational weeks. This study will fill a gap in human milk research in China, provide theoretical basis for the superiority of breastfeeding, and provide more powerful nutritional support for the catch-up growth of preterm infants

DETAILED DESCRIPTION:
Objective:

1. Analyze and compare the differences in HMOs components among mothers who give birth at different gestational weeks;
2. Longitudinal observation of weekly changes in HMOs concentrations of premature mothers within 1 month of delivery;
3. Validate the association between HMOs components in preterm mothers and fecal intestinal flora in infants at 6 months of age.

Research content

1. The LC-MS method will be used to detect the content of HMOs in preterm mothers and compared with the corresponding components in term breast milk during the postpartum period to analyze the effects of different gestational weeks on HMOs;
2. The intestinal flora 16S rDNA high-throughput sequencing method will be used to determine the bacterial gene profile in the fecal DNA samples of infants, and the differences between the gestational age groups (term and preterm infants) were compared, and the preterm infants in this group were plotted Evolution of intestinal flora within 6 months of birth;
3. Use statistical methods to verify the association between HMOs components in preterm mothers and the establishment of intestinal flora in infants.

ELIGIBILITY:
Inclusion Criteria:

* (1) Be healthy, have no acute or chronic diseases, have no severe complications during pregnancy
* (2) Breastfeeding for more than 6 months and Volunteer to participate in this study (signed informed consent)
* (3) Age of maternal women: 20~35years
* (4) Breast milk is sufficient, and the amount of milk secreted each time is more than 30ml
* (5) No fatal, important organ system deformities and metabolic defects in neonates

Exclusion Criteria:

* (1) for infants: Rescued to death or hospitalized due to critical illness during the study period
* (2)for lactating mothers: exposure to tobacco and alcohol during lactation, severe postpartum depression and other mental and psychological diseases, obesity (BMI> 28), use of antibiotics or antimetabolites, mastitis with fever within 7 days before specimen collection (T> 38.5 ℃),Suspension or termination of breastfeeding in the state of maternal and infant illness

Ages: 7 Days to 35 Years | Sex: All
Age Groups: Child, Adult
Study Population: Lactating mothers and infants in cooperative maternity hospital
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2019-04-08 (Actual); Primary Completion 2021-10 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Human milk oligosaccharide detection | Day7-12, Day14-19, Day21-26, Day28-33
  Liquid chromatography-mass spectrometer(LC-MS) will be used to quantitatively detect a total of 15 types of neutral oligosaccharides and acid oligosaccharides in different breast milk samples.
  Human milk samples will be collected four times for each mother after delivery (day7-12, day14-19, day21-26, day28-33). Only one series of samples will be collected for each mother, and 30 samples are needed for each group, totaling 480 human milk samples

SECONDARY OUTCOMES:
To dectect the intestinal flora with16s RNA high throughput sequencing | Day7-12, Day28-33, 3 months and 6 months
  The results of bacterial gene profiles in fecal DNA samples of premature infants at different gestational ages will be analyzed as follows.First, bacterial genomic DNA in feces will be obtained using the QIAamp Fast DNA Stool Mini Kit(51604), and PCR amplification will be performed. After the Miseq library are successfully constructed, cluster preparation and sequencing will be performed with qualified libraries. The data obtained by the machine will be used for biological information analysis. By comparing OTU with database, species annotation will be performed on OTU.Based on OTU and species annotation results, species complexity analysis and inter-group species difference analysis will be carried out.
  Neonatal fecal samples will be collected four times for each infant after delivery at day7-12, day28-33, 3 months and 6 months of age. Only one series of samples will be collected from each infant, and 30 samples are needed for each group, totaling 480 fecal samples.
Achieved the body weight of infants | Day7-12, Day14-19, Day21-26, Day28-33, 2 months, 3 months, 4months and 6 months.
  Measured the body weight (grams) of infants at 8 time points: Day7-Day12, Day14-Day19, Day21-Day26, Day28-Day33, 2 months, 3 months, 4months and 6 months.
Achieved the body length of infants | Day7-12, Day14-19, Day21-26, Day28-33, 2 months, 3 months, 4months and 6 months.
  Measured the body length (mm) of infants at 8 time points: Day7-Day12, Day14-Day19, Day21-Day26, Day28-Day33, 2 months, 3 months, 4months and 6 months.
Achieved the head circumference of infants | Day7-12, Day14-19, Day21-26, Day28-33, 2 months, 3 months, 4months and 6 months.
  Measured the head circumference (mm) of infants at 8 time points: Day7-Day12, Day14-Day19, Day21-Day26, Day28-Day33, 2 months, 3 months, 4months and 6 months.
Stool status of infants | Day7-12, Day14-19, Day21-26, Day28-33, 2 months, 3 months, 4months and 6 months.
  Achieved the stool status( frequency, color, character)of neonatal based on health consultation at 8 time points: Day7-Day12, Day14-Day19, Day21-Day26, Day28-Day33, 2 months, 3 months, 4months and 6 months.
Average daily formula intake | Day7-12, Day14-19, Day21-26, Day28-33, 2 months, 3 months, 4months and 6 months.
  Achieved the average daily formula intake volume at 8 time points: Day7-Day12, Day14-Day19, Day21-Day26, Day28-Day33, 2 months, 3 months, 4months and 6 months.
Disease and medication history | 6 months
  Record the disease and medication history of infants in each group

CONTACTS AND LOCATIONS:
Overall Officials: Jing Li, PhD, Principal Investigator — Shanghai Children's Medical Center
Locations (1):
- Shanghai first maternal and infant health care hospital, Shanghai, China